CLINICAL TRIAL: NCT01575730
Title: Phase II Study Comparing Normothermic Versus Hyperthermic Intraoperative Chemoperfusion With Oxaliplatin in Patients With Peritoneal Metastases From Appendiceal or Colon Cancer
Brief Title: Cytoreduction Followed by Normothermic Versus Hyperthermic Intraperitoneal Intraoperative Chemoperfusion (HIPEC): a Study in Peritoneal Carcinomatosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/237; 2012-000701-77 (EudraCT Number)
Record Dates: First submitted 2012-04-06; First posted 2012-04-11 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Peritoneal Carcinomatosis
Keywords: Peritoneal carcinomatosis from colorectal or appendiceal origin
MeSH Terms: conditions — Peritoneal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oxaliplatin 37°C, high dose, 30 minutes (Active Comparator)
  Interventions: Procedure: Hyperthermic intraoperative Peritoneal Chemoperfusion
- Oxaliplatin 41 °C, high dose, 30 minutes (Placebo Comparator)
  Interventions: Procedure: Hyperthermic intraoperative Peritoneal Chemoperfusion
- Oxaliplatin 37°C, low dose, 90 minutes (Active Comparator)
  Interventions: Drug: Hyperthermic intraoperative Peritoneal Chemoperfusion

INTERVENTIONS:
Procedure: Hyperthermic intraoperative Peritoneal Chemoperfusion — Dose: 460 mg/m², duration: 30 minutes, temperature 37°C
  Arms: Oxaliplatin 37°C, high dose, 30 minutes
Procedure: Hyperthermic intraoperative Peritoneal Chemoperfusion — Dose: 460 mg/m², duration: 30 minutes, temperature 41°C
  Arms: Oxaliplatin 41 °C, high dose, 30 minutes
Drug: Hyperthermic intraoperative Peritoneal Chemoperfusion — Dose: 200 mg/m², duration: 90 minutes, temperature 37°C
  Arms: Oxaliplatin 37°C, low dose, 90 minutes

SUMMARY:
Peritoneal carcinomatosis from appendix or colon (large bowel) cancer is treated in suitable patients with surgery followed by instillation of heated chemotherapy inside the abdominal cavity. This procedure is termed 'Hyperthermic intraoperative Peritoneal Chemoperfusion' or HIPEC. Many center perform HIPEC with high dose oxaliplatin, a standard chemotherapy drug active against colon cancer, administered during 30 minutes at 41°C. The hypothesis of this study is, that chemoperfusion at normal (37.5°C) temperature but longer duration (90 minutes) may be safer and at least as efficient. Patients will be treated with one of three possible HIPEC regimens using oxaliplatin: high dose, 30 min, 41°C; high dose, 30 min, 37.5°C; or low dose, 90 min, 37.5°C. The outcome parameters are pharmacokinetic and pharmacodynamic: using specialized techniques, tissue penetration of chemotherapy and cancer cell kill effects will be compared in order to establish the safest and most active HIPEC regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peritoneal carcinomatosis from colorectal origin (including appendiceal mucinous neoplasms and the pseudomyxoma syndromes) amenable for cytoreduction and HIPEC.

Exclusion Criteria:

* No written informed consent
* Irresectable and/or metastatic disease found during surgery
* Known allergy to oxaliplatin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-05-21 (Actual); Primary Completion 2013-03-18 (Actual); Study Completion 2013-03-18 (Actual)

PRIMARY OUTCOMES:
Morbidity | Until discharge or within 30 days
  Scoring of postoperative morbidity according to the Dindo-Clavien system
Mortality | Until discharge or within 30 days
  The number of deaths will be recorded.
Area under the perfusate concentration versus time curve (AUC) of platinum | Before addition of chemotherapy, at 10, 20 and 30 minutes after addition of chemotherapy
  Measurements of platinum in perfusate samples on the high dose interventions.
Area under the perfusate concentration versus time curve (AUC) of platinum | Before addition of chemotherapy, at 10, 20, 30, 40, 50, 60, 70, 80 and 90 minutes after addition of chemotherapy
  Measurements of platinum in perfusate samples on the low dose intervention.
Area under the plasma concentration versus time curve (AUC) of platinum | Before addition of chemotherapy, at 10, 20, 30,45, 60, 90 minutes and 2, 4, 8, 12, 18, 24 hours after addition of chemotherapy
  Measurements of platinum in perfusate samples on the high dose interventions.
Area under the plasma concentration versus time curve (AUC) of platinum | Before addition of chemotherapy, at 10, 20, 30, 40, 50, 60, 70, 80, 90 minutes and 2, 4, 8, 12, 18, 24 hours after addition of chemotherapy
  Measurements of platinum in plasma samples on the low dose intervention.

SECONDARY OUTCOMES:
Tissue Concentration (Cmax) of Platinum | after 30 or 90 minutes
  Platinum concentration will be measured after removal of perfusate.

CONTACTS AND LOCATIONS:
Overall Officials: Wim P Ceelen, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be